CLINICAL TRIAL: NCT00533429
Title: Protocol H6Q-MC-S034(a) Randomized, Double-Blind, Phase 2 Study of Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin Versus Pemetrexed + Carboplatin + Bevacizumab + Placebo in Chemonaive Patients With Stage IIIB or IV Non-Small Cell Lung Cancer
Brief Title: Study of Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin Versus Pemetrexed + Carboplatin + Bevacizumab + Placebo in Participants With Non-Small Cell Lung Cancer Who Have Not Been Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11398; H6Q-MC-S034 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — enzastaurin; Pemetrexed; Carboplatin; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin
  Interventions: Drug: enzastaurin; Drug: pemetrexed; Drug: carboplatin; Drug: bevacizumab
- B (Placebo Comparator): Pemetrexed + Carboplatin + Bevacizumab + Placebo
  Interventions: Drug: pemetrexed; Drug: carboplatin; Drug: bevacizumab; Drug: Placebo

INTERVENTIONS:
Drug: enzastaurin — 1125 milligram (mg) loading dose then 500 mg, oral, daily until disease progression
  Other Names: LY317615
  Arms: A
Drug: pemetrexed — 500 milligrams per square meter (mg/m^2), intravenously ( IV), Day 8 of cycle 1 - 28 days, Day 1 of subsequent cycles every (q) 21 days x 3 cycles
  Other Names: LY231514; Alimta
Drug: carboplatin — Area under the curve (AUC) 6, IV, Day 8 cycle 1 - 28 days, Day 1 of subsequent cycles q 21 days x 3 cycles
Drug: bevacizumab — 15 milligrams/kilogram (mg/kg), IV, Day 8 of cycle 1 - 28 days, Day 1 of subsequent cycles q 21 days x 3 cycles
Drug: Placebo — oral, daily
  Arms: B

SUMMARY:
The purpose of this study is to determine if Pemetrexed plus Carboplatin plus Bevacizumab plus Enzastaurin, followed by maintenance Bevacizumab plus Enzastaurin can extend survival time without disease progression in the first-line treatment of participants with advanced stage non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* participants or their legal representative must have signed an informed consent document for clinical research
* have laboratory confirmed diagnosis of advanced, nonsquamous cell non-small cell lung cancer (NSCLC) (Stage IIIB or IV disease) which is not curable
* have not received any prior systemic chemotherapy, immunotherapy, targeted therapy, or biological therapy for advanced NSCLC, prior radiation therapy is allowed to less than 25% of the bone marrow
* have measurable disease
* have adequate organ function and estimated life expectancy of 12 weeks

Exclusion Criteria:

* have known central nervous system (CNS) disease; major surgery within 28 days; minor surgery within 7 days; serious concomitant systemic disorder; serious cardiac condition; have a serious, nonhealing wound, ulcer, or bone fracture
* have received treatment within the last 30 days with any drug that has not received regulatory approval for any indication at the time of study entry
* have previously received treatment with enzastaurin, pemetrexed, or bevacizumab
* are pregnant or breast-feeding
* are unable to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bentonville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galesburg, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomington, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Muncie, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow reports those participants who discontinued from study drug.
Groups:
- Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin: Combination biochemotherapy:
  Pemetrexed: 500 milligrams per square meter (mg/m^2) intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Carboplatin: Area under the curve (AUC) 6 intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Bevacizumab: 15 milligrams/kilogram (mg/kg) intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Enzastaurin: 1125 milligram (mg) loading dose on Day 1 of Cycle 1 (28 days), followed by 500 mg oral daily dose for 3 cycles
  Maintenance therapy:
  Enzastaurin: 500 mg oral daily dose for 21-day cycles until disease progression
  Bevacizumab: 15 mg/kg intravenously on Day 1 of every 21-day cycle until disease progression
- Pemetrexed + Carboplatin + Bevacizumab + Placebo: Combination biochemotherapy:
  Pemetrexed: 500 mg/m^2 intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Carboplatin: AUC 6 intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Bevacizumab: 15 mg/kg intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Placebo: Oral tablets daily to complete Cycle 1 (28 days), then subsequent 21-day cycles for 3 cycles
  Maintenance therapy:
  Bevacizumab: 15 mg/kg intravenously on Day 1 of every 21-day cycle until disease progression
  Placebo: Oral tablets daily for 21-day cycles until progressive disease
Period: Overall Study
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin | Pemetrexed + Carboplatin + Bevacizumab + Placebo
Started | 20 | 20
Received at Least 1 Dose of Study Drug | 20 | 20
Entered Maintenance | 8 | 10
Completed | 1 | 4
Not Completed | 19 | 16
Not completed — Adverse Event | 3 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Progressive Disease | 12 | 13
Not completed — Symptomatic deterioration | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin | Pemetrexed + Carboplatin + Bevacizumab + Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.3) | 61.2 (9.0) | 61.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status classifies participants according to their functional impairment.
  Participants
    0 - Fully Active | 10 | 11 | 21
    1 - Ambulatory, Restricted Strenuous Activity | 10 | 9 | 19
Prior therapy [Count of Participants; unit: Participants] — Prior therapy included radiation, surgery and chemotherapy in an adjuvant setting.
  Participants
    Yes | 3 | 3 | 6
    No | 17 | 17 | 34
Disease Stage [Count of Participants; unit: Participants] — Cancer staging is a process describing the severity of the cancer, size of the tumor and how far it has spread from the original location. Stage IIIB: a tumor of any size that has spread (metastasized) to distant lymph nodes, has invaded other structures in the chest (such as the heart or esophagus), or has a malignant pleural effusion (fluid build-up containing cancer cells between the layers lining the lungs). Stage IV: a tumor of any size that has spread (metastasized) to another region of the body or to another lobe of the lungs.
  Participants
    Stage IIIB | 3 | 3 | 6
    Stage IV | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from date of randomization to the first observation of progressive disease (PD) or death due to any cause. For participants not known to have died as of the data cutoff date and who did not have objective PD, PFS was censored at the date of the last objective progression-free assessment. For participants who received subsequent anticancer therapy (after discontinuation from all study treatment) prior to objective disease progression or death, PFS was censored at the date of the last objective progression-free assessment prior to the initiation of post-discontinuation anticancer therapy.
Time Frame: Randomization to measured PD or death from any cause up to 12.2 months
Population: All randomized participants identified by assigned treatment group. Number of participants censored: Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin = 5; Pemetrexed + Carboplatin + Bevacizumab + Placebo = 2.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin | Pemetrexed + Carboplatin + Bevacizumab + Placebo
Number analyzed (Participants) | 15 | 18
months | 3.5 [2.0 to 5.8] | 4.3 [2.5 to 5.8]
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin vs Pemetrexed + Carboplatin + Bevacizumab + Placebo; Test type: Superiority or Other; p = 0.469, Log Rank — P-value (one-tailed) was calculated based on the un-stratified log-rank test

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Response Rate)
Description: Tumor response rate was defined as number of participants with overall best response of CR or PR over number of protocol qualified participants using the Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria. CR was defined as the disappearance of all tumor lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum of LDs or complete disappearance of target lesions, with persistence (but not worsening) of 1 or more non-target lesions. In either case, no new lesions may have appeared.
  Percentage of participants was calculated as: (number of participants with CR or PR/ number of participants qualified for tumor response analysis) × 100.
Time Frame: Randomization to measured progressive disease or death from any cause up to 12.2 months
Population: All randomized participants identified by assigned treatment group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin | Pemetrexed + Carboplatin + Bevacizumab + Placebo
Number analyzed (Participants) | 20 | 20
percentage of participants | 20.0 [2.5 to 37.5] | 30.0 [9.9 to 50.1]
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin vs Pemetrexed + Carboplatin + Bevacizumab + Placebo; Test type: Superiority or Other; p = 0.462, Fisher Exact — 95% confidence interval based on normal approximation to the binomial distribution. P-value (2-tailed) calculation based on unadjusted, normal-distribution approximation for the difference in rates

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. For participants who were not known to have died as of the data cutoff, OS was censored at the last contact date.
Time Frame: Randomization to date of death up to 14.3 months
Population: All randomized participants identified by assigned treatment group. Participants censored: Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin = 12; Pemetrexed + Carboplatin + Bevacizumab + Placebo = 9.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin | Pemetrexed + Carboplatin + Bevacizumab + Placebo
Number analyzed (Participants) | 8 | 11
months | 9.1 [7.8 to NA] — Not calculable due to high number of censored participants. | 7.6 [4.2 to NA] — Not calculable due to high number of censored participants.
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin vs Pemetrexed + Carboplatin + Bevacizumab + Placebo; Test type: Superiority or Other; p = 0.492, Log Rank — P-value (two-tailed) was calculated based on the un-stratified log-rank test

4. Secondary Outcome: Time to Progressive Disease (TTPD)
Description: TTPD was defined as the time from the date of randomization until the first date of objectively determined progressive disease (PD). For participants who died without objective PD (including death from study disease), TTPD was censored at the date of the last objective progression-free disease assessment. For participants not known to have died as of the data cutoff and did not have PD, TTPD was censored at the date of the last objective progression-free disease assessment.
Time Frame: Randomization to measured PD or death from any cause up to 12.2 months
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Enzastaurin + Pemetrexed + Carboplatin + Bevacizumab: Combination biochemotherapy:
  Pemetrexed: 500 milligrams per square meter (mg/m^2) intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Carboplatin: Area under the curve (AUC) 6 intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Bevacizumab: 15 milligrams/kilogram (mg/kg) intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Enzastaurin: 1125 milligram (mg) loading dose on Day 1 of Cycle 1 (28 days), followed by 500 mg oral daily dose for 3 cycles
  Maintenance therapy:
  Enzastaurin: 500 mg oral daily dose for 21-day cycles until disease progression
  Bevacizumab: 15 mg/kg intravenously on Day 1 of every 21-day cycle until disease progression
Arm/Group | Enzastaurin + Pemetrexed + Carboplatin + Bevacizumab | Pemetrexed + Carboplatin + Bevacizumab + Placebo
Number analyzed (Participants) | 20 | 20
Months | 4.3 [1.7 to 5.8] | 4.8 [3.0 to 7.2]

5. Secondary Outcome: Duration of Response (DoR)
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death from any cause. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST v1.0) criteria. CR was defined as the disappearance of all target lesions and PR was defined as having at least a 30% decrease in sum of longest diameter (LD) of target lesions taking as reference the baseline sum of LDs. For participants who died without progressive disease or who were alive, DoR was censored at the last contact of progression free assessment. For participants who received subsequent anticancer therapy (after discontinuation from all study treatment) prior to PD, DoR was censored at the date of last progression-free assessment prior to the initiation of post-discontinuation anticancer therapy. Due to early study closure, DoR was not analyzed.
Time Frame: Time of response to disease progression or death from any cause up to 12.2 months
Population: All randomized participants. Participants censored: Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin = 16; Pemetrexed + Carboplatin + Bevacizumab + Placebo = 14.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin | Pemetrexed + Carboplatin + Bevacizumab + Placebo
Number analyzed (Participants) | 4 | 6
Months | 4.7 [2.8 to NA] — The upper 95% confidence interval was not achieved due to high censoring rate. | 3.5 [1.3 to NA] — The upper 95% confidence interval was not achieved due to high censoring rate.

6. Secondary Outcome: Pharmacology Toxicity and Adverse Events (AEs)
Description: Clinically significant events were defined as serious AEs (SAEs) and other non-serious AEs. Participants who died due to progressive disease (PD) or an AE while on treatment and or died during the 30 day post-treatment follow-up are included. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Randomization up to 14.3 months and 30-day follow-up
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Pemetrexed + Carboplatin + Bevacizumab + Placebo: Combination biochemotherapy:
  Pemetrexed: 500 mg/m^2 intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Carboplatin: AUC 6 intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Bevacizumab: 15 mg/kg intravenously on Day 8 of Cycle 1 (28 days), then on Day 1 of subsequent cycles every 21 days for 3 cycles
  Placebo: Oral tablets daily to complete Cycle 1 (28 days), then subsequent 21-day cycles for 3 cycles
  Maintenance therapy:
  Bevacizumab: 15 mg/kg intravenously on Day 1 of every 21-day cycles until disease progression
  Placebo: Oral tablets daily for 21-day cycles until progressive
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin | Pemetrexed + Carboplatin + Bevacizumab + Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Non-serious AEs | 19 | 20
  Serious AEs | 6 | 7
  Deaths Due to PD | 0 | 0
  Deaths Due to AEs | 1 | 1
  Deaths within 30-days after treatment | 0 | 0

ADVERSE EVENTS:
Time Frame: Randomization up to 14.3 months and 30-day follow-up
Description: Study-specific clinical outcomes due to progressive disease were not considered to be a serious adverse event (SAE) unless the investigator deemed it related to the use of the study drug.
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin | Pemetrexed + Carboplatin + Bevacizumab + Placebo
Serious Adverse Events (participants affected / at risk) | 6/20 | 7/20
Other Adverse Events (participants affected / at risk) | 19/20 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin (N=20) | Pemetrexed + Carboplatin + Bevacizumab + Placebo (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Confusional state (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pemetrexed + Carboplatin + Bevacizumab + Enzastaurin (N=20) | Pemetrexed + Carboplatin + Bevacizumab + Placebo (N=20)
Leukopenia (Blood and lymphatic system disorders) | 13 (32) | 14 (53)
Lymphopenia (Blood and lymphatic system disorders) | 5 (9) | 2 (12)
Eye disorder (Eye disorders) | 0 (0) | 2 (2)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 10 (12) | 9 (12)
Diarrhoea (Gastrointestinal disorders) | 6 (15) | 7 (9)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (19) | 10 (16)
Peritoneal infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (7) | 9 (11)
Fatigue (General disorders) | 16 (32) | 12 (37)
Hyperhidrosis (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 2 (4) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Urticaria (Immune system disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Pelvic infection (Infections and infestations) | 1/9 (1) | 0/10 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 6 (14)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 7 (12)
Blood alkaline phosphatase increased (Investigations) | 5 (9) | 5 (5)
Blood creatinine increased (Investigations) | 3 (5) | 2 (5)
Ear, nose and throat examination abnormal (Investigations) | 8 (13) | 4 (5)
Haemoglobin decreased (Investigations) | 17 (51) | 18 (58)
Neutrophil count decreased (Investigations) | 10 (21) | 10 (39)
Platelet count decreased (Investigations) | 13 (33) | 15 (48)
Weight decreased (Investigations) | 3 (4) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 11 (13) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (7) | 3 (7)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (7) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (8) | 4 (4)
Hypothyroidism (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (3)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Confusional state (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 5 (6)
Insomnia (Nervous system disorders) | 6 (8) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (4) | 1 (2)
Depression (Psychiatric disorders) | 3 (5) | 2 (3)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Hot flush (Reproductive system and breast disorders) | 1/9 (1) | 0/10 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 6 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dizziness (Vascular disorders) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 9 (10) | 5 (6)
Haemorrhage (Vascular disorders) | 0 (0) | 3 (4)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Respiratory tract haemorrhage (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days